CLINICAL TRIAL: NCT06488456
Title: Psychometric Properties of the Turkish Version of Therapy-Related Symptom Checklist for Children Scale
Brief Title: Psychometric Properties of the Therapy-Related Symptom Checklist-Children
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, SEDA ARDAHAN SEVGİLİ, Assistant Professor, Ege University
Other Study IDs: 22-3.1T/16
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Leukemia, Acute Myeloid; Pediatric ALL
Keywords: psychometric properties; symptom; pediatrics; nursing care
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: TRSC-C — Data were collected using TRSC-C

SUMMARY:
Diagnosis and treatment of childhood cancers is an exhausting process that affects both children and their caring parents physically and mentally. While the survival rate in childhood cancers was 28% in the 1960s, this rate has increased up to 80% with the developments in treatment methods. Although the main methods used in cancer treatment today are surgical treatment, radiotherapy, and immunotherapy, the main component of cancer treatment is chemotherapy. Improvements in chemotherapy protocols have increased survival; however, the use of high-dose chemotherapy may increase the frequency and severity of symptoms that may be seen in children. Therefore, diagnosis and management of treatment-related symptoms in the pediatric population receiving chemotherapy treatment as soon as possible is of vital importance as it will significantly affect the quality of life of children. In this context, this study aimed to add to the national literature by conducting a Turkish validity and reliability study of a checklist suitable for the use of health professionals in clinics for monitoring the side effects of chemotherapy. In the study, validity and reliability tests will be performed for intercultural scale adaptation.

DETAILED DESCRIPTION:
Leukaemias are the most common type of cancer in children and young people, accounting for 1/3 of all cancers in the population. Most childhood leukaemias are acute lymphocytic leukaemia (ALL), while the rest of the cases are acute myeloid leukaemia (AML). In childhood, ALL peaks at the age of 2-4 years. AML, on the other hand, can be seen throughout childhood and is more common in children under 2 years of age and in adolescents. Chronic leukaemias are rarely seen in children.

After the leukaemia is diagnosed and the type of leukaemia is determined, the treatment protocol is decided according to the risk group of the disease. The main treatment for childhood leukaemia is chemotherapy. For children in the high-risk group, high-dose chemotherapy may be given together with stem cell transplantation. Treatment of leukaemias can last 2-3 years with maintenance treatment, depending on the type and risk group. Chemotherapy is known to cause many side effects in both adults and children. The most well-known of these side effects are nausea and vomiting, loss of appetite, weight loss, mucositis, gastrointestinal system changes and fatigue, alopecia, pain, depression.

Monitoring and effective management of side effects of chemotherapy is one of the most important aspects of cancer treatment. Symptoms resulting from the use of chemotherapies require careful monitoring to identify adverse side effects on patients. During the diagnosis and treatment process of leukaemia, children experience many symptoms at the same time. When these symptoms are both related to each other and occur at the same time, this is called a symptom cluster. Studies emphasise that multiple symptoms are seen in children and adolescents with cancer. When the literature was analysed, it was seen that there were few studies involving the use of checklists to identify symptoms and symptom management, the sample of which consisted of patients and their parents in Turkey. However, recognising symptom clusters may provide a better understanding of the structure of multiple symptoms and more effective symptom management. In this context, this study aimed to add to the national literature by conducting a Turkish validity and reliability study of a checklist suitable for the use of health professionals in clinics for monitoring the side effects of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 2-18 years of age
* The patient has received chemotherapy treatment at least twice,
* The patient/caregiver parent speaks Turkish and is open to communication
* Volunteering to participate in the study.

Exclusion Criteria:

* The patient is younger than 2 years of age
* The patient has never received chemotherapy
* The subject/caregiver parent does not speak Turkish
* The patient is being treated for a disease other than leukemia

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 2-18 who are receiving chemotherapy treatment for leukaemia in the relevant clinic/polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Turkish version of the scale | April 2022-December 2024
  Use of the Turkish version of the Theraphy Related Symptom Checklist. Min: 0, Max: 120 points The higher the score, the worse the symptoms.

SECONDARY OUTCOMES:
frequency of symptoms | April 2022-December 2024
  frequency of symptoms related to chemotherapy treatment
symptom severity | April 2022-December 2024
  symptom severity due to chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seda Ardahan Sevgili, PhD, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study data are not shared due to ethical rules and laws. If necessary, it will be shared with the relevant parties if requested